CLINICAL TRIAL: NCT04866056
Title: A Multicentric Phase I/II Study of Jaktinib Hydrochloride Tablets in Combination With Azacitidine for Injection in Patients With Myelodysplastic Syndromes(MDS) With Myelofibrosis(MF) or MDS/Myeloproliferative Neoplasms With MF
Brief Title: Jaktinib and Azacitidine In Treating Patients With MDS With MF or MDS/MPN With MF.
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Corporate policy adjustments
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZGJAK019
Record Dates: First submitted 2021-04-28; First posted 2021-04-29 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Myelodysplastic Syndromes; Myeloproliferative Neoplasms; Myelofibrosis
Keywords: MDS; MF; MPN
MeSH Terms: conditions — Myelodysplastic Syndromes; Myeloproliferative Disorders; Primary Myelofibrosis | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment(Jaktinib+Azacitidine) (Experimental): Patients receive azacitidine subcutaneously (SC) on days 1-7 and Jaktinib orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Jaktinib; Drug: azacitidine

INTERVENTIONS:
Drug: Jaktinib — Jaktinib PO BID
Drug: azacitidine — Azacytidine SC

SUMMARY:
This phase I/II trial studies how well Jaktinib and azacytidine work in treating patients with myelodysplastic syndromes with myelofibrosis or myelodysplastic syndrome/myeloproliferative neoplasm with myelofibrosis. Giving Jaktinib and azacytidine may be an effective treatment for myelodysplastic syndromes with myelofibrosis or myelodysplastic syndrome/myeloproliferative neoplasm with myelofibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily sign the informed consent form (ICF);
* Age ≥ 18 years, either male or female;
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
* Expected life expectancy is greater than 24 weeks;
* Diagnosis of myelodysplastic syndrome/myeloproliferative neoplasm (MDS/MPN) according to World Health Organization (WHO)；
* The patients understands the purpose of and procedures required for the study and is willing to participate in the study；

Exclusion Criteria:

* Subjects with congestive heart failure, uncontrolled or unstable angina or myocardial infarction,cerebrovascular accident, or pulmonary embolism within 6 months prior to screening;
* Subjects suffering from arrhythmia and requiring treatment, or QTcB > 480ms at screening;
* Subjects with clinical symptoms of active bacterial, viral, parasitic or fungal infections requiring treatment at screening;
* Subjects with known human immunodeficiency virus (HIV), known active infectious Hepatitis B (HepB), and/or known active infectious Hepatitis C (HepC);
* Female subjects who are pregnant, currently breastfeeding, planning to become pregnant;
* Subjects who had experienced malignant tumors (except for adequately treated local basal cell or squamous cell carcinoma of the skin and cervical carcinoma in situ that have been cured) within the past 5 years;
* Subjects who have any other conditions that are not specified in the protocol but the investigator believes that they are not suitable for inclusion in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Objective response rate (complete remission+partial remission+marrow compete remission +cytogenetic complete remission + hematological improvement) in patients with Myelodysplastic Syndromes | Up to16 weeks
  According to the 2006 International Working Group (IWG) response criteria in myelodysplasia，The objective response rate will be estimated along with the Bayesian 95% credible interval.
Objective response rate (complete remission+cytogenetic complete remission+partial remission+clinical improvement) in patients with myelodysplastic syndromes/myeloproliferative neoplasms | Up to16 weeks
  According to the 2015 ICP in MDS/MPN. The objective response rate will be estimated along with the Bayesian 95% credible interval.

SECONDARY OUTCOMES:
Overall survival | Time from treatment start till death or last follow-up, assessed up to 2 years
  Will be listed and summarized by the Kaplan-Meier estimator
Duration of response | Duration from the first documented onset of partial response or complete response to the date of progressive disease/relapse, assessed up to 2 years
  Will be listed and summarized by the Kaplan-Meier estimator
Relapse-free survival | Time from start of response to the date of event defined as the first documented progressive disease/relapse or death, whichever comes first, assessed up to 2 years
  Will be listed and summarized by the Kaplan-Meier estimator

CONTACTS AND LOCATIONS:
Locations (1):
- 79 Qingchun Road, Hangzhou, Zhejiang, China